CLINICAL TRIAL: NCT00441090
Title: A Phase 2 Double-Blind, Randomized, Dose-Ranging, Placebo-Controlled, Parallel Group Study of AKR-501 Tablets Taken Orally Once Daily for 28 Days in Patients With Chronic Idiopathic Thrombocytopenic Purpura (ITP).
Brief Title: Study of AKR-501 Tablets Taken Orally Once Daily for 28 Days in Patients With Chronic Idiopathic Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AKR-501-CL-003
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Chronic Idiopathic Thrombocytopenic Purpura; Purpura, Thrombocytopenic, Idiopathic
Keywords: Chronic Idiopathic Thrombocytopenic Purpura; Idiopathic Thrombocytopenic Purpura; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avatrombopag tablets (Experimental): 2.5, 5, 10 or 20 mg tablets
  1 tablet taken orally once daily for 28 days
  Interventions: Drug: Avatrombopag tablets
- Placebo tablet (Placebo Comparator): 2.5, 5, 10, or 20 mg tablets
  1 tablet taken orally once daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo tablets 2.5, 5, 10 and 20 mg taken orally once daily for 28 days.
  Arms: Placebo tablet
Drug: Avatrombopag tablets — Avatrombopag tablets 2.5, 5, 10 and 20 mg taken orally once daily for 28 days.
  Other Names: AKR-501; E5501; YM477
  Arms: Avatrombopag tablets

SUMMARY:
The purpose of this study is to determine the efficacy, safety and tolerability, of AKR-501 (avatrombopag) tablets, as compared to placebo, in the treatment of participants with chronic Idiopathic Thrombocytopenic Purpura (ITP).

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, double-blind, randomized, placebo-controlled, dose-ranging, parallel-group study. The pharmacokinetic (PK) and pharmacokinetic/pharmacodynamic (PK/PD) relationship of avatrombopag will also be studied. Approximately 65 eligible participants will be randomized in a 3:3:3:3:1 ratio in a double-blinded fashion into one of five parallel treatment groups to receive daily doses of either avatrombopag 2.5, 5, 10 or 20 mg or placebo for 28 days, respectively. Each avatrombopag dosing group will consist of 15 participants while the placebo group will consist of 5 participants. All study participants will be evaluated weekly (Days 3, 5, 7, 14, 21 and 28) for safety, efficacy, and (Days 7, 14, 21, and 28) avatrombopag PK while receiving study treatment with a final assessment for safety and effectiveness to be done 2 weeks after the last study dose (Day 42).

At the completion of Visit Day 28±1, participants who complete 28±1 days of study dosing will be assessed for eligibility to enroll into the rollover Study 501-CL-004 (NCT00625443) based on this visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Confirmed diagnosis of ITP according to American Society of Hematology (ASH) Guidelines ≥ 3 months prior to Day 1.
3. If ≥ 60 years old, must have had either a bone marrow biopsy consistent with ITP within past 3 years or a good response (platelet count > 100,000/mm^3) to a previous ITP treatment.
4. Are refractory or relapsed after at least one prior ITP therapy (patients who are refractory and failed to achieve a platelet count ≥ 50,000/mm^3 despite steroids or ≥ 30,000/mm^3 to other prior ITP therapies, such as splenectomy, danazol, or immunosuppressive drugs. For patients who are relapsed, the platelet counts must be below 50,000/mm^3 if using steroids or 30,000/mm^3 if not prescribed steroids.)
5. Patients receiving maintenance corticosteroids may be enrolled, as long as the corticosteroids have been administered at a stable dose (same milligram amount ± 10%) for ≥ 2 weeks prior to Screening Visit A and the investigator does not foresee the need to change the steroid dose during study participation. Patients should remain on this stable corticosteroid dose during study participation.
6. Patients receiving stable dosages of cyclosporine A, mycophenolate mofetil, azathioprine or danazol may also be enrolled. The dosages of all these medications must be stable for at least 3 months prior to AKR-501 administration.
7. Platelet count:

   * Patients not receiving steroids (no steroid treatment for > 2 weeks prior to the Screening Visit A): platelets < 30,000/mm^3 at Screening Visit A and within 96 hours prior to Day 1 (Screening Visit B)
   * Patients receiving steroids: platelets < 50,000/mm^3 at Screening Visit A and within 96 hours prior to Day 1 (Screening Visit B).
8. Women of child-bearing potential must have a negative pregnancy test at Screening Visit A and Screening Visit B. (Childbearing potential is defined as any woman who has not been surgically sterilized and is premenopausal or peri-menopausal i.e., any menstrual flow within 12 months of Screening Visit A).
9. Women of child-bearing potential and all men must agree to practice a medically approved form of contraception (one of the following must be used: condoms (male or female) with a spermicidal agent, diaphragm, or cervical cap with a spermicidal agent, IUD, hormonal contraception, abstinence).
10. Willing and able to provide written informed consent before any study-related procedure.

Exclusion Criteria:

1. Women who are pregnant and/or lactating.
2. Splenectomy procedure performed 4 weeks prior to AKR-501 administration.
3. Use of the following drugs or treatments prior to Day 1:

   * Within 3 months - Rituximab;
   * Within 2 weeks - Aspirin or Aspirin-containing compounds, Salicylates, Anticoagulants, clopidogrel, ticlopidine, Rh0(D) Immune Globulin (WinRho®), or intravenous immunoglobulin (IVIG).
4. Participation in a clinical trial involving any investigational agent within 4 weeks of Day 1.
5. Exposure to eltrombopag or AMG -531.
6. Significant medical conditions or diseases as determined by the Investigator (e.g., clinically active systemic lupus erythematosus; known or suspected HIV infection; acute hepatitis or clinically active chronic hepatitis; lymphoproliferative disease; congestive heart failure).
7. History of cardiovascular disease (e.g., angina, unstable angina, myocardial infraction, coronary artery stent placement, angioplasty, coronary artery bypass grafting).
8. History of thromboembolic disease (e.g., transient ischemic attack [TIA], stroke [CVA], pulmonary embolism [PE]).
9. History of deep venous thrombosis (DVT).
10. History of lupus anticoagulant or anticardiolipin antibody syndrome or positive anti b2 glycoprotein antibody.
11. History of any medical condition where systemic anticoagulation was required for more than 6 months.
12. Laboratory abnormalities:

    * Hemoglobin < 12.5 g/dL for men and < 11.5 g/dL for women. If anemia is clearly related to ITP, for example excessive blood loss, then that patient may be enrolled without the need for a waiver after discussion with the Sponsor's medical monitor
    * White blood cell count (WBC) < lower limit of normal
    * Absolute neutrophil count (ANC) < 1000/mm^3
    * Prothrombin time (PT) > 1.25 x upper limit of normal
    * Partial thromboplastin time (PTT) > 1.25 x upper limit of normal
    * Total bilirubin > 3 x upper normal limit
    * Alanine transaminase (ALT) > 3 x upper normal limit
    * Aspartate transaminase (AST) > 3 x upper normal limit
    * Creatinine > 1.5x upper normal limit
    * Blood urea nitrogen (BUN) > 1.5 x upper normal limit
    * HIV positive
    * IgM HAV positive, Hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV) positive.
13. History of, or current alcohol or drug abuse likely to interfere with ability to comply with protocol.

    requirements or give informed consent, as determined by the Investigator.
14. History of, or current psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent, as determined by the Investigator.
15. Currently taking any of the following medications: Rituximab, Aspirin or Aspirin-containing compounds, Salicylates, Anticoagulants, clopidogrel, ticlopidine, Rh0(D) Immune Globulin (WinRho®), or intravenous immunoglobulin (IVIG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ran Ho, MD, Study Director — Eisai Inc.
Locations (25):
- United States (25):
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Bay Area Cancer Research Group, LLC, Concord, California
  - Pacific Coast Hematology/Oncology Medical Group Inc., Fountain Valley, California
  - University of California Irvine Cancer Center, Orange, California
  - Davis, Posteraro and Wasser, MDs, LLP, Manchester, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Florida Cancer Institute, New Port Richey, Florida
  - Columbus Clinic, PC, Columbus, Georgia
  - John H. Stroger, Jr. Hospital of Cook County, Div. of Hematology and Oncology, Chicago, Illinois
  - Comprehensive Bleeding Disorders Center, Peoria, Illinois
  - Cancer Care Center, Inc., New Albany, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Kansas City Cancer Center, LLC, Kansas City, Missouri
  - UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - New York Presbyterian Hospital, Weill Medical College of Cornell University, New York, New York
  - Emerywood Oncology and Hematology, High Point, North Carolina
  - Mid Ohio Oncology/Hematology, Inc., dba The Mark H. Zangmeister Center, Columbus, Ohio
  - UPENN, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolina, Greenville, South Carolina
  - Puget Sound Blood Center, Seattle, Washington

REFERENCES:
- [Derived] Bussel JB, Kuter DJ, Aledort LM, Kessler CM, Cuker A, Pendergrass KB, Tang S, McIntosh J. A randomized trial of avatrombopag, an investigational thrombopoietin-receptor agonist, in persistent and chronic immune thrombocytopenia. Blood. 2014 Jun 19;123(25):3887-94. doi: 10.1182/blood-2013-07-514398. Epub 2014 May 6. PMID 24802775

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.5 mg Avatrombopag: 2.5 mg tablet taken orally once daily for 28 days
- 5.0 mg Avatrombopag: 5.0 mg tablet taken orally once daily for 28 days
- 10.0 mg Avatrombopag: 10.0 mg tablet taken orally once daily for 28 days
- 20.0 mg Avatrombopag: 20.0 mg tablet taken orally once daily for 28 days
- Placebo: 3:3:3:3:1 ratio to avatrombopag tablet taken orally once daily for 28 days
Period: Overall Study
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo
Started | 15 | 15 | 14 | 15 | 5
Completed | 13 | 14 | 12 | 13 | 5
Not Completed | 2 | 1 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Platelet increase;more than 500,000 mm^3 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized (Intent-to-Treat) population included all participants who were randomly assigned to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 5 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (17.84) | 55.6 (18.03) | 57.5 (17.88) | 47.9 (16.54) | 39.6 (20.63) | 52.3 (17.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 8 | 11 | 3 | 40
  Male | 6 | 6 | 6 | 4 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate (RR) to Avatrombopag on Day 28
Description: Platelet counts were measured from the participant's blood, which was drawn at their Screening Visit B (Day -4 to Day 1, Baseline), and on study drug treatment Day 28. The RR was defined as the percentage of participants with a Day 1 platelet count of less than 30,000/milliliter (mL) who reached a platelet count of greater than or equal to 50,000/mL on Day 28 of study medication, together with the percentage of participants using steroids who had a Day 1 platelet count greater than or equal to 30,000/mL but less than 50,000/mL who reached a platelet count of greater than or equal to 20,000/mL higher than their Day 1 platelet count on Day 28 of study medication. The RR was summarized by treatment group using the method of last observation carried forward (LOCF).
Time Frame: Day-4 to Day 1, Baseline, Day 28
Population: Full analysis population, LOCF, included participants who were randomly assigned to treatment and had at least one post-baseline platelet count assessment. The randomized, full analysis, and safety populations were identical for this study. No participants were excluded from the efficacy analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 5
Percentage of participants | 13.3 | 53.3 | 50.0 | 80.0 | 0

2. Secondary Outcome: Change in Platelet Count From Baseline
Description: Platelet counts were measured from the participant's, blood which was drawn at their Screening Visit B (Day -4 to Day 1, Baseline), and on study drug treatment Days 7, 14, 21, and 28. The unit of measure was "K/mm^3", where "K = platelets x 1000 = platelets x 10^3" and "mm^3 = cubic milliliter= microliter".
Time Frame: Day -4 to Day 1, Baseline, Day 7, Day 14, Day 21, Day 28
Population: Full Analysis population, LOCF
Measure: Mean (Standard Deviation); unit: platelets x 10^3/mm^3
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 5
platelets x 10^3/mm^3
  Day 7 | 13.6 (22.37) | 46.7 (55.22) | 68.3 (81.23) | 168.8 (114.59) | 5.0 (9.54)
  Day 14 | 12.5 (22.64) | 57.5 (74.72) | 103.1 (119.55) | 332.4 (278.96) | -1.4 (4.16)
  Day 21 | 7.5 (18.38) | 47.1 (54.54) | 80.6 (129.98) | 261.3 (278.17) | 8.4 (13.72)
  Day 28 | 7.3 (23.74) | 43.7 (50.35) | 81.0 (124.55) | 200.2 (292.36) | -1.8 (7.73)

3. Secondary Outcome: Responder Rate to Avatrombopag by Visit
Description: Platelet counts were measured from the participant's blood, which was drawn at their Screening Visit B (Day -4 to Day 1, Baseline), and on study drug treatment Days 7, 14, and 21. The RR was summarized by treatment group using the method of LOCF. Day 28 was not included with this data because it was reported as a primary outcome measure.
Time Frame: Day -4 to Day 1, Baseline, Day 7, Day 14, and Day 21
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 5
Percentage of participants
  Day 7 | 6.7 | 66.7 | 64.3 | 93.3 | 0
  Day 14 | 20.0 | 60.0 | 78.6 | 93.3 | 0
  Day 21 | 13.3 | 60.0 | 50.0 | 86.7 | 0

4. Secondary Outcome: Percentage of Participants With Platelet Counts Greater Than or Equal to 50,000/mL by Visit
Description: Platelet counts were measured from the participant's blood, which was drawn at their Screening Visit B (Day -4 to Day 1, Baseline), and on study drug treatment Days 7, 14, 21, and 28.
Time Frame: Day -4 to Day 1, Baseline, Day 7, Day 14, Day 21, and Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 5
Percentage of participants
  Day 7 | 6.7 | 66.7 | 64.3 | 93.3 | 0
  Day 14 | 20.0 | 60.0 | 78.6 | 93.3 | 0
  Day 21 | 13.3 | 60.0 | 50.0 | 86.7 | 20.0
  Day 28 | 13.3 | 53.3 | 50.0 | 80.0 | 0

5. Secondary Outcome: Percentage of Participants With Platelet Counts Greater Than or Equal to 100,000/mL by Visit
Description: Platelet counts were measured from the participant's, blood which was drawn at their Screening Visit B (Day -4 to Day 1, Baseline), and on study drug treatment Days 7, 14, 21, and 28.
Time Frame: Day -4 to Day 1, Baseline, Day 7, Day 14, Day 21, and Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 5
Percentage of participants
  Day 7 | 6.7 | 20.0 | 28.6 | 80.0 | 0
  Day 14 | 0 | 26.7 | 42.9 | 86.7 | 0
  Day 21 | 0 | 20.0 | 21.4 | 73.3 | 0
  Day 28 | 6.7 | 33.3 | 28.6 | 53.3 | 0

6. Secondary Outcome: Percentage of Participants Whose Platelet Counts Doubled From Baseline by Visit
Description: as for outcome 5
Time Frame: Day -4 to Day 1, Baseline, Day 7, Day 14, Day 21, and Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 5
Percentage of participants
  Day 7 | 33.3 | 60.0 | 78.6 | 93.3 | 20.0
  Day 14 | 26.7 | 60.0 | 71.4 | 93.3 | 0
  Day 21 | 6.7 | 60.0 | 64.3 | 86.7 | 20.0
  Day 28 | 13.3 | 53.3 | 57.1 | 86.7 | 20.0

7. Other Pre Specified Outcome: To Evaluate the Pharmacokinetics (PK) and the Pharmacokinetic/Pharmacodynamic (PK/PD) Relationship of Avatrombopag in Patients With ITP.
Description: Given the sparse PK sampling in this study, PK data from outside studies, which includes healthy subjects, were included to assist in PK model development. As a result this data was not reported with these study results.
Time Frame: Days 7, 14, 21 and 28
Population: Given the sparse PK sampling in this study, PK data from outside studies, which includes healthy subjects, were included to assist in PK model development. As a result this data was not reported with these study results.
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from first dose of study drug until last follow-up visit, or 30 days following discontinuation of study drug, whichever occurred later, or approximately 91 days.
Description: Safety population included all participants who received at least one dose of study drug and had at least one safety assessment. Treatment-emergent AEs and SAEs are new events, or worsening of pre-existing events, that occur after the first dose of study drug and were reported in this section.
Arm/Group | 2.5 mg Avatrombopag | 5.0 mg Avatrombopag | 10.0 mg Avatrombopag | 20.0 mg Avatrombopag | Placebo
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/15 | 1/14 | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 12/15 | 13/15 | 11/14 | 14/15 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2.5 mg Avatrombopag (N=15) | 5.0 mg Avatrombopag (N=15) | 10.0 mg Avatrombopag (N=14) | 20.0 mg Avatrombopag (N=15) | Placebo (N=5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Renal artery occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 0
Gastric haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2.5 mg Avatrombopag (N=15) | 5.0 mg Avatrombopag (N=15) | 10.0 mg Avatrombopag (N=14) | 20.0 mg Avatrombopag (N=15) | Placebo (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Tympanic membrance disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Auricular swelling (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal upper pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral mucosal petechiae (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Bowel sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 4 | 4 | 2 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 0
Hunger (General disorders) | 0 | 0 | 0 | 1 | 0
Mucosal haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Furnuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Horeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngtis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 4 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 1 | 4 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Anxiety (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Vasoconstriction (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other